CLINICAL TRIAL: NCT02409927
Title: Effect of Medium-chain Triglycerides Emulsification on Ketogenesis and Adverse Effects in Human Adults
Brief Title: Effect of MCT Emulsification on Ketogenesis in Human Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-391
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Medium-chain triglycerides; Metabolism; Ketones; Lipids; Emulsification
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Each participant underwent 7 metabolic day (1-day visit), each visit separate by a minimum of 3 day
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy participant (Other): Each participant undergo 7 metabolic day, separate by at least 3 days, where they received a different dietary supplement on each day: control (no supplement), MCT oil 10g, MCT oil 20g, MCT oil 30g (provided from pure MCT oil), MCT homogenate 10g, MCT homogenate 20g, MCT homogenate 30g (provided by a 10% MCT homogenate emulsion)
  Interventions: Dietary Supplement: MCT oil 10g; Dietary Supplement: MCT homogenate 10g; Dietary Supplement: Control; Dietary Supplement: MCT oil 20g; Dietary Supplement: MCT homogenate 20g; Dietary Supplement: MCT oil 30g; Dietary Supplement: MCT homogenate 30g

INTERVENTIONS:
Dietary Supplement: MCT oil 10g — 10 g of pure MCT oil mixed with skim milk in a standardized breakfast
Dietary Supplement: MCT homogenate 10g — 10g provided by 10% MCT homogenate mixed with skim milk in a standardized breakfast
Dietary Supplement: Control — vehicule (skim milk) with a standardized breakfast
Dietary Supplement: MCT oil 20g — 20g of pure MCT oil mixed with skim milk in a standardized breakfast
Dietary Supplement: MCT homogenate 20g — 20g provided by 10% MCT homogenate mixed with skim milk in a standardized breakfast
Dietary Supplement: MCT oil 30g — 30g of 100% pure MCT oil mixed with skim milk in a standardized breakfast
Dietary Supplement: MCT homogenate 30g — 30g provided by 10% MCT homogenate mixed with skim milk in a standardized breakfast

SUMMARY:
Lower brain glucose uptake is present before the onset of cognitive deterioration and may increase the risk of cognitive decline in Alzheimer's disease. Ketones are the brain's main alternative energy substrates. Medium-chain triglycerides (MCT) are rapidly beta-oxidized and are ketogenic. Large doses of MCT oil are linked to gastro-intestinal side effects due to incomplete absorption so the investigators examined whether homogenisation into a skim milk matrix (MCT-H) would both improve ketogenesis and reduce side-effects compared to MCT taken without homogenisation into a matrix (bulk MCT [MCT-B]).

Hypotheses: (i) MCT-H will be better absorbed compared to MCT-B, so MCT-H will result in higher ketonemia and lower side effects in healthy adults. (ii) The effects of MCT-B and MCT-H on ketogenesis will be dose-dependent.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or more

Exclusion Criteria:

* smoker
* pregnancy or breastfeeding
* diabetes or insulin resistance
* uncontrolled thyroid disease, hepatic or renal disease
* uncontrolled high blood pressure
* medical treatment influencing lipid or glucide metabolism
* ongoing or past severe drug or alcohol abuse
* dementia or psychiatric difficulties or depression
* chronic immune condition or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen C Cunnane, PhD, Principal Investigator — Université de Sherbrooke

REFERENCES:
- [Derived] Courchesne-Loyer A, Lowry CM, St-Pierre V, Vandenberghe C, Fortier M, Castellano CA, Wagner JR, Cunnane SC. Emulsification Increases the Acute Ketogenic Effect and Bioavailability of Medium-Chain Triglycerides in Humans: Protein, Carbohydrate, and Fat Metabolism. Curr Dev Nutr. 2017 Jun 21;1(7):e000851. doi: 10.3945/cdn.117.000851. eCollection 2017 Jul. PMID 29955713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Participant
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy: Participants involved in the project had seven metabolic study day to do : control day (no supplement), MCT oil 10,20 or 30 g, and MCT homogenate 10, 20 or 30 g. They were taking the supplement with a breakfast and there was blood sampling every 30 minutes.t
Arm/Group | Healthy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 31 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Plasma Ketone Concentration
Description: Average of total ketones (beta-hydroxynutyrate + acetoacetate) measured in plasma, measured every 30 minutes for hours following intake of the different supplements
Time Frame: Average of every 30 minutes for 4 hours following intake of supplement
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Healthy Participant
Number analyzed (Participants) | 10
µmol/L
  control | 136.97 (11.33)
  10g MCT oil | 177.43 (14.711)
  20 g MCT oil | 270.61 (27.477)
  30 g MCT oil | 249.3 (17.474)
  10g MCT homogenate | 262.92 (26.82)
  20g MCT homogenate | 277.25 (30.006)
  30 g MCT homogenate | 244.74 (65.83)

2. Secondary Outcome: Plasma Glucose Concentration
Description: average of glucose measured every 30 minutes during the four hour of each metabolic day
Time Frame: Average of every 30 minutes for 4 hours following intake of supplement
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Healthy Participant
Number analyzed (Participants) | 10
mmol/L
  control | 4.86 (0.33)
  10 g MCT oil | 4.98 (0.24)
  20g MCT oil | 4.97 (0.28)
  30g MCT oil | 4.99 (0.27)
  10g MCT homogenate | 5.01 (0.26)
  20g MCT homogenate | 4.84 (0.26)
  30g MCT homogenate | 5.09 (0.22)

3. Secondary Outcome: Plasma Free Fatty Acids Concentration
Description: average of free fatty acids measured every 30 minutes during the four hour fo each metabolic day
Time Frame: average of 4 hours following intake of supplement
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Healthy Participant
Number analyzed (Participants) | 10
µmol/L
  control | 0.43 (0.05)
  10g MCT oil | 0.39 (0.04)
  20g MCT oil | 0.41 (0.04)
  30 g MCT oil | 0.38 (0.05)
  10g MCT homogenate | 0.44 (0.05)
  20g MCT homogeante | 0.41 (0.05)
  30g MCT homogenate | 0.5 (0.06)

4. Secondary Outcome: Plasma Insuline Concentration
Description: Average of insulin measured evey 30 minutes during the 4 hours of each metabolic day
Time Frame: average of 4 hours following intake of supplement
Measure: Mean (Standard Error); unit: µIU/mL
Arm/Group | Healthy Participant
Number analyzed (Participants) | 10
µIU/mL
  control | 9.79 (2.03)
  10g MCT oil | 13.7 (3.43)
  20 g MCT oil | 10.88 (2.01)
  30 g MCT oil | 13.00 (2.58)
  10g MCT homogenate | 12.87 (2.47)
  20g MCT homogenate | 11.94 (2.84)
  30g MCT homogenate | 12.86 (2.08)

5. Secondary Outcome: Number of Participants With Side Effects for Each Visit
Description: If participant had any side effect (mild or moderate) at least one time during the day.
Time Frame: During the 4 hours following intake of supplement
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participant
Number analyzed (Participants) | 10
Participants
  control | 0
  10 g MCT oil | 1
  20 g MCT oil | 4
  30 g MCT oil | 5
  10 g MCT homogenate | 2
  20g MCT homogenate | 4
  30g MCT homogenate | 5

ADVERSE EVENTS:
Time Frame: Adverse event date were collected during the 7 metabolic study day
Arm/Group | Healthy Participant
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Participant (N=10)
Abnominal discomfort (Gastrointestinal disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
gastric reflux (Gastrointestinal disorders) | 2
Nausea (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 0
Headache (General disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes